CLINICAL TRIAL: NCT05977855
Title: Use of a Diary to Assess and Monitor Behavioral and Psychological Symptoms of Dementia
Brief Title: Use of a Diary to Assess and Monitor Behavioral and Psychological Symptoms of Dementia ( BPSDiary )
Acronym: BPSDiary
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS San Gerardo dei Tintori (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPSDiary
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Behavioral and Psychiatric Symptoms of Dementia
Keywords: Behavioral and Psychiatric Symptoms of Dementia; Randomized Clinical Trial; Diary
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diary (Experimental)
  Interventions: Other: BPSDiary
- Standard Care (No Intervention)

INTERVENTIONS:
Other: BPSDiary — The BPSDiary is a diary to register severity, hour, day and triggers of a number of BPSD (namely, agitation, aggression, delusions/hallucinations, insomnia, aberrant motor behavior).
  Arms: Diary

SUMMARY:
The goal of this randomized clinical trial is to compare the efficacy of the use of a diary to record behavioral and psychological symptoms of dementia (BPSD) in persons with dementia. The main questions it aims to answer are:

* Does the use of a diary lead to a reduction of the caregiver's burden at 3 months, compared with standard care?
* Does the use of a diary lead to a reduction of the neuropsychiatric inventory (NPI) score at 3 months, compared with standard care?
* Does the use of a diary result in less psychotropic drugs prescribed to the patient at 3 months compared with standard care?
* Are physicians and caregivers satisfied with managing patients with the use of a diary?
* Does the use of a diary reduce the caregiver's stress related to BPSD at 3 months, compared with standard care? Participants will be randomly assigned to either the use of a diary or a control group. Caregivers in the diary arm will be asked to fill in a diary with BPSD including triggers, severity, day and hour, to be analyzed by physicians to prescribe appropriate pharmacological or non-pharmacological interventions. The control group will receive usual care (i.e., appropriate interventions will be applied after interviewing the caregiver and/or visiting the patient).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cognitive impairment (neurodegenerative or vascular)
* Caregiver and patient willing to participate in the study
* Caregiver living with the patient or able to cover all 24 hours
* Presence of BPSD pertaining to the hyperactivity-irritability-impulsivity-disinhibition cluster (HIDA)
* Signed informed consent before the beginning of the study

Exclusion Criteria:

* Refusal to consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Zarit Burden Interview | 3 months
  Zarit Burden Interview difference between intervention arm and controls

SECONDARY OUTCOMES:
Neuropsychiatric Inventory | 3 months
  Neuropsychiatric Inventory difference between intervention arm and controls
Olanzapine equivalents | 3 months
  Calculated with the Defined Daily Doses method; difference between intervention arm and controls
Satisfaction questionnaire | 3 months
  A questionnaire to evaluate care-related satisfaction in caregivers and physicians (range 0-32, higher scores indicate better outcomes); difference between intervention arm and controls
Neuropsychiatric Inventory - Caregiver Distress Scale | 3 months
  Subscale of NPI-caregiver distress scale relative to the domains included in the diary (range 0-35, higher scores indicate worse outcomes); difference between intervention arm and controls

CONTACTS AND LOCATIONS:
Locations (9):
- Italy (9):
  - Ospedale SS Annunziata, Chieti, Abruzzo
  - Pia Fondazione Card. Panico, Tricase, Apulia
  - Università Sapienza, Rome, Lazio
  - Ospedale Multimedica, Castellanza, Lombardy
  - Fondazione IRCCS Don Gnocchi, Milan, Lombardy
  - Fondazione IRCCS San Gerardo dei Tintori [Recruiting], Monza, Lombardy
  - Fondazione IRCCS Mondino, Pavia, Lombardy
  - AOU Careggi, Florence, Tuscany
  - AO Padova, Padua, Veneto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pozzi FE, Cali L, D'Antonio F, Altomare AI, Sepe Monti M, Panigutti M, Di Crosta A, Palumbo R, Bonanni L, Carlucci V, Busse C, Cagning A, Urso D, Vilella D, Logroscino G, Alberoni M, Bellinvia A, Farina E, de Rino F, Gavazzi A, Zuffi M, Bruno G, Bessi V, Cotta Ramusino M, Perini G, Costa A, Ferrarese C, Appollonio I, Tremolizzo L. BPSDiary study protocol: a multi-center randomized controlled trial to compare the efficacy of a BPSD diary vs. standard care in reducing caregiver's burden. Front Dement. 2023 Dec 18;2:1301280. doi: 10.3389/frdem.2023.1301280. eCollection 2023. PMID 39081982